CLINICAL TRIAL: NCT07096726
Title: Boston Medical Center Ultrasound Decongestion Study
Brief Title: Boston Medical Center Ultrasound Decongestion Study in Heart Failure
Acronym: BUDS-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-44593
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Congestive Heart Failure; Volume Overload
Keywords: Venous Excess Ultrasound (VExUS); Ultrasound-assisted diuresis; Heart Failure with Preserved Ejection Fraction (HFpEF); Heart Failure with Reduced Ejection Fraction (HFrEF)
MeSH Terms: conditions — Heart Failure; Edema | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants in the emergency department, on the floors, or in the outpatient heart failure infusion clinic will be randomly allocated in a 1:1 ratio to the study arms.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants in both arms will be blinded as they will receive VExUS scan throughout their admission. For the control arm, the treatment team (clinicians) will be blinded to the VExUS scores and will conduct SOC with the patient for the course of their admission. All investigator sonographers performing the VExUS scans will be blinded to arm assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Five-point ultrasound guided diuresis (Experimental): Participants randomized to this study arm will have their diuresis guided by five-point ultrasound to assess venous congestion and receive standard of care.
  Interventions: Device: Five-point ultrasound; Other: Standard of care
- Standard of care guided diuresis (Active Comparator): Participants randomized to this study arm will have their diuresis clinically guided by standard of care. They will also have five point ultrasound but the results will not inform their diuresis.
  Interventions: Device: Five-point ultrasound; Other: Standard of care

INTERVENTIONS:
Device: Five-point ultrasound — In-person study visits will be done on initial evaluation and then at least every 48 hours, during which serial five-point ultrasound will be performed to assess venous congestion. Each visit will not be at strict intervals; a reasonable time window is every 48 hours +/- 12 hours. Ultrasound may be performed more frequently if clinically indicated. During these visits or between them, ultrasound of the heart may additionally be performed. Each visit will last between 10 and 60 minutes.
Other: Standard of care — Standard of care will most likely include radiographic investigations (chest X-ray, chest CT), laboratory evaluation (complete blood counts, metabolic panel, B-type natriuretic peptide, high-sensitivity troponin, electrolytes, renal function, urine testing), volume status, and cardiopulmonary physical exam.

SUMMARY:
The purpose of this study is to analyze the utility of a novel five-point ultrasound as a predictor of volume overload in diverse patients who are admitted with volume overload/congestive heart failure (CHF) exacerbation at Boston Medical Center (BMC), the largest safety-net hospital in New England. Current standard of care (SOC) involves the utilization of laboratory markers and physical exam, which is often inconsistent and equivocal. The investigators will assess will assess if ultrasound-assisted diuresis reduces recurrent episodes of volume overload/decompensated heart failure.

DETAILED DESCRIPTION:
This superiority randomized clinical trial will compare the therapeutic intervention of five-point ultrasound-guided diuresis with standard of care diuresis for decompensated heart failure. Participants with heart failure exacerbation will be randomly allocated in a 1:1 ratio using heart failure patient lists, by a heart failure physician in the emergency department or on the floors. Similarly, patients will be randomly selected in a 1:1 ratio in the outpatient heart failure infusion clinic when seen for heart failure exacerbation by a heart failure physician. The study population will be generally stable and can be inpatient or outpatient.

The primary objective of the study is to evaluate and compare the efficacy of diuresis when driven by standard of care or five-point ultrasound to guide clinical decision making by assessing 30-day hospital readmission rate in patients undergoing standard of care vs ultrasound assisted diuresis.

The specific aims are:

Aim 1. To measure and compare changes in ultrasonographic parameters (ultrasound Doppler profiles, VExUS scores) through the course of a HF hospitalization for decongestion for acute decompensated HF admission.

Aim 2. To compare 30-day and 90-day HF readmission rates between randomized patients with HF admission comparing SOC to VExUS-guided decongestion strategy.

Aim 3: To compare worsening renal failure/acute renal injury (defined as 25% increase in serum Cr/cystatin C from time of admission to 4 weeks post-discharge) between randomized admitted HF patients comparing SOC to VExUS-guided decongestion strategy.

Secondary objectives include:

1. To assess differences in diuretic responsiveness in individuals with varying cardiac dysfunction (i.e., length of stay for patients with HFpEF vs HFrEF)
2. To assess differences in diuretic responsiveness in individuals with varying right ventricular function
3. To assess differences in hospital length of stay between SOC and VExUS-guided decongestion groups
4. To assess differences in 30- and 90-day mortality between SOC and VExUS-guided decongestion groups
5. To assess differences in need for renal replacement therapy between SOC and VExUS-guided decongestion groups

ELIGIBILITY:
Inclusion Criteria:

* Patient with a primary diagnosis of acute on chronic decompensated heart failure who is admitted to inpatient or presents to the outpatient Boston Medical Center (BMC) Heart Failure Infusion clinic for decongestion treatment.
* Willing and able to receive short abdominal and thoracic ultrasounds throughout hospitalization
* Patients with right and/or left ventricular failure

Exclusion Criteria:

* Hemodynamic instability defined as systolic blood pressure <85 mmHg or mean arterial pressure <60 mm Hg for greater than 24 hours duration
* Abdominal surgery in the past 1 month
* Significant acute or chronic liver disease
* End stage renal disease on dialysis
* Advanced chronic kidney disease (CKD) [Stage V CKD with glomerular filtration rate (GFR) <15] to exclude renal vein doppler ultrasound
* Severe acute kidney injury (AKI) or requiring renal replacement therapy
* Known abdominal thrombus in the inferior vena cava (IVC) or portal vein
* Acute myocarditis
* Acute valvular disease
* Acute type 1 myocardial infarction
* Medical condition precluding abdominal ultrasound due to significant discomfort or pain
* Adults not able to provide consent (a simple teach back method of key aspects discussed in consent form will be utilized to verify if patient is able to adequately provide informed consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
VExUS Doppler profiles and scores | At admission, At discharge (on average 3-10 days)
  The range of VExUS profiles and scores to guide clinicians with heart failure diuresis are: No congestion (normal inferior vena cava), Minimal congestion (0 or 1 abnormal doppler patterns). Mild congestion (2 abnormal patterns and portal vein pulsatility fraction [PVPF] less than 30%), Moderate congestion (2 abnormal patterns and PVPF between 30 and 50%), Severe congestion (2 abnormal patterns and PVPF more than 50%).
30-day hospital readmission rate | 30 days after discharge (on average 3-10 days)
  The number of any hospital readmissions within 30 days of discharge will be abstracted from the participants' electronic medical records.
90-day hospital readmission rate | 90 days after discharge (on average 3-10 days)
  The number of any hospital readmissions within 90 days of discharge will be abstracted from the participants' electronic medical records.
Worsening renal failure/acute renal injury | admission to 4 weeks post discharge (on average 3-10 days)
  This outcome is defined by an increase in 25% of serum creatinine or serum cystatin C from the time of admission to 4 weeks post discharge. It will be abstracted from the participants' electronic medical records.

SECONDARY OUTCOMES:
Hospital length-of-stay for decompensated heart failure | At hospital discharge (on average 3-10 days)
  The total number of days hospitalized for decompensated heart failure will be abstracted from the participants' electronic medical records.
30-day HF readmission rate | 30 days post discharge (on average 3-10 days)
  The number of readmissions within 30-days of hospital discharge that are specifically due to HF
All-cause mortality | 30 days, 90 days
  All-cause mortality will be abstracted from the participants' electronic medical records.
Need for renal replacement therapy | 30 days, 90 days
  The need for renal replacement therapy will be abstracted from the participants' electronic medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Deepa M Gopal, MD, Principal Investigator — Boston Medical Center, Cardiovascular Medicine/Heart Failure; Aala Jaberi, MD, Principal Investigator — Boston Medical Center, Nephrology Section
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No